CLINICAL TRIAL: NCT06066996
Title: Evaluation of the Electronic Cigarette Withdrawal Syndrome: Mechanistic Targets for Intervention
Brief Title: Evaluation of the Electronic Cigarette Withdrawal Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00407275; R01DA057925 (NIH)
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: E-cigarette Use; Withdrawal
MeSH Terms: conditions — Vaping | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Transdermal Nicotine Patch (Experimental): Participants assigned to this condition will receive a blinded nicotine patch and will wear the patch on their upper arm, per the manufacturer's instructions.
  Interventions: Drug: Transdermal Nicotine Patch
- Transdermal Placebo Patch (Placebo Comparator): Participants assigned to this placebo nicotine patch condition will receive a blinded patch containing 0mg of nicotine, and will wear the patch on their upper arm, per the manufacturer's instructions.
  Interventions: Drug: Placebo Nicotine Patch
- No Patch (No Intervention): Participants assigned to this condition will not receive a patch.

INTERVENTIONS:
Drug: Transdermal Nicotine Patch — Blinded Nicotine Patch
  Arms: Transdermal Nicotine Patch
Drug: Placebo Nicotine Patch — Blinded Patch with No Nicotine
  Arms: Transdermal Placebo Patch

SUMMARY:
The goal of this project is to rigorously evaluate the nature of e-cigarette withdrawal in exclusive e-cigarette users during a monitored abstinence period and the role of nicotine in the expression of this withdrawal syndrome.

DETAILED DESCRIPTION:
This project will use a rigorous residential laboratory design to evaluate e-cigarette withdrawal expression and experimentally determine the role of nicotine in this syndrome. Healthy adults who exclusively use e-cigarettes will undergo monitored e-cigarette abstinence over seven days (1 week) in a residential unit. The investigators will evaluate the contribution of nicotine to withdrawal expression by assigning participants to one of three conditions: active nicotine patch, placebo patch control, or no patch to control for expectancies. Standardized behavioral and biological measures associated with withdrawal including patient report, cognitive task performance, and biometrics will be collected throughout to establish a rigorous timecourse of withdrawal and evaluate the contribution of nicotine to these symptoms.

ELIGIBILITY:
Inclusion criteria:

1. 21-55 years old
2. good general health as reviewed by study medical team
3. vital signs in normal range as reviewed by study medical team
4. negative urine test for illicit drug use (excluding THC) and negative breath alcohol test
5. daily use of a nicotine-containing e-cigarette for at least 6 months
6. no regular use of other tobacco products (e.g., smokeless products) for at least 6 months
7. urine cotinine >100ng/mL (i.e., recommended cutoff for confirming current nicotine use)
8. exhaled breath carbon monoxide (CO) <6ppm
9. Penn State E-cigarette Dependence (PSED) score >=4, indicating mild dependence or greater
10. have an interest in reducing e-cigarette use

Exclusion criteria:

1. psychoactive drug use (aside from cannabis, nicotine, alcohol, caffeine) in past month
2. current use of over-the-counter (OTC) or prescription medications that may impact safety
3. use cannabis >2 times per week
4. history of or current significant medical condition that would impact participation or safety according to the study investigators and medical staff
5. current psychiatric condition or substance use disorder (aside from tobacco use disorder) that would impact participation or safety according to the study investigators and medical staff
6. enrollment in another trial
7. positive pregnancy test
8. currently using a nicotine/tobacco cessation product
9. seizure disorder or traumatic brain injury (TBI)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hughes-Hatsukami Withdrawal Scale | Baseline, every 4 hours up to 16 hours
  The Hughes-Hatsukami Withdrawal Scale consists of 13 items presented individually on a 100mm visual analog scale. Higher scores reflect higher withdrawal (worse outcome) [range 0-32]. Measures are taken at baseline, 8am, 12pm, 4pm, and 8pm every day during the seven day residential stay.
Change in Smoking urges as assessed by the Tiffany-Drobes Questionnaire of Smoking Urges (QSU) Brief | Baseline, every 4 hours up to 16 hours
  The Tiffany-Drobes QSU Brief consists of ten items, each presented on the screen as a phrase centered above seven boxes ranging from (strongly disagree) to (strongly agree). Higher scores reflect higher withdrawal (worse outcome) [range 0-70]. Measures are taken at baseline, 8am, 12pm, 4pm, and 8pm every day during the seven day residential stay.
Change in Positive and Negative Affect Schedule (PANAS) | Baseline, every 4 hours up to 16 hours
  The PANAS consists of 20 items presented individually on a five-point Likert scale. Higher scores reflect more positive affect and negative affect [range 0-50]. Measures are taken at baseline, 8am, 12pm, 4pm, and 8pm every day during the seven day residential stay.
Change in Conners' Continuous Performance Task (CPT) | Baseline, every 4 hours up to 16 hours
  On the CPT, participants respond to single letters appearing on their computer screen but are asked to refrain from responding to a specified letter(i.e., the letter X). Higher scores reflect more inattention. Measures are taken at baseline, 8am, 12pm, 4pm, and 8pm every day during the seven day residential stay.
Change in Memory as assessed by the N-Back | Baseline, every 4 hours up to 16 hours
  On the n-back, participants decide whether each stimulus in a sequence matches the one that appeared "n" items ago. Higher scores reflect more accuracy. Measures are taken at baseline, 8am, 12pm, 4pm, and 8pm every day during the seven day residential stay.
Total sleep time | Nightly up to seven days
  Total time sleeping in minutes measured using actigraphy and unobtrusive EEG.
Total time spent in Rapid eye movement (REM) sleep | Nightly up to seven days
  Total time sleeping in minutes in REM stage measured using actigraphy and unobtrusive EEG.
Wake after sleep onset (WASO) | Nightly up to seven days
  Total number of minutes that a person is awake after having initially fallen asleep measured using actigraphy and unobtrusive EEG.

SECONDARY OUTCOMES:
Change in E-Cigarette Demand Intensity | Baseline, every 4 hours up to 16 hours
  E-cigarette use at unconstrained price measured using a commodity purchase task. Higher scores reflect more demand (worse outcome). Measures are taken at baseline, 8am, 12pm, 4pm, and 8pm every day during the seven day residential stay.
Change in E-Cigarette Demand Elasticity | Baseline, every 4 hours up to 16 hours
  Sensitivity of e-cigarette use to price measured using a commodity purchase task. Higher scores reflect more price sensitivity (better outcome). Measures are taken at baseline, 8am, 12pm, 4pm, and 8pm every day during the seven day residential stay.
Return to Use | Day 14
  Return to e-cigarette use at the one week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Strickland, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States